CLINICAL TRIAL: NCT02616536
Title: Comparison Between Traditional Classroom Teaching Verses Flipped Classroom Teaching on Knowledge Gain of Physiotherapy Students
Brief Title: Comparison Between Teaching Methods on Knowledge Gain of Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Manisha Parai, Lecturer, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UniversitiTAR
Record Dates: First submitted 2015-11-19; First posted 2015-11-30 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Educational Activities
Keywords: Flipped classroom; Teaching methods; Knowledge gain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flipped classroom (Active Comparator): The flipped classroom is new pedagogical method, which employs asynchronous video lectures and practice problems as homework and active, group-based problem solving activities in the classroom.
  Interventions: Other: Teaching methods
- traditional classroom (Active Comparator): The classroom lecture is a special form of communication in which voive, gesture. Movements, facial expression and eye contact can either complement or detract from the content. No matter what your topic, your delivery and manner of speaking immeasurably influence your student's' attentiveness and learning.
  Interventions: Other: Teaching methods

INTERVENTIONS:
Other: Teaching methods — the two teaching methods will be given to two groups of students and their knowledge gain will be analysed

SUMMARY:
Procedures:

The study will be conducted in two phases:

Phase 1

* Perception and Satisfaction questionnaire will be developed
* A validation test will be conducted on the Perception and Satisfaction questionnaire (face, content and construct) before conducting the study. The validation process will involve the participation of lecturers, professors and students by convenience sampling.

Phase 2

* To prevent bias from the researchers, each participant will be given their code as their identification number. Then the participants will be randomly divided into two groups. They will be briefed on the purpose of study (stating that, the investigators would like to see the efficacy of various teaching methods on students' knowledge gain) and procedure of the study (examinations will be conducted, surveys at the end of each class session and at the end of the study). They are requested to fill up basic demographic data, consent form and ILS questionnaire(measuring the learning style of student) before beginning the study.
* In this study, the lecture will be given by the 'Researcher 1' to standardize the input to the participants of the two groups. This will produce a standardized input to the students of the two groups of teaching method.
* For the FC (flipped classroom) group, the length of the pre-recorded lecture videos will be the same which the participants can view it unlimitedly. An assignment will be given for FC group that will be attempted during the discussion class(2 hours) a week after with the lecturer. No grades will be given for the assignment.
* Meanwhile for the TC(traditional classroom) group, a standard lecture class of 1 hour and 1 hour of tutorial class will be conducted on the same topic. The same ungraded assignment will also be given to this group a week after the lecture class to be attempted in the tutorial class
* One day gap will be given following the discussion and tutorial class for FC and TC groups respectively following which an examination of 1 hour duration will be conducted to test on their level of knowledge (assessed by exam score) on the topic being taught for both the groups using the same set of questions.
* At the end of the study, each participant will be given a feedback questionnaire to evaluate their perception and satisfaction on the teaching method applied on them using the 'Perception and Satisfaction Questionnaire'.

DETAILED DESCRIPTION:
Study Design:

Effectiveness of flipped classroom compared to traditional lecture classroom among physiotherapy participants - Quasi Experimental Study: This method of study divides a group of participants from respective year and semester into two groups, controlled (traditional lecture) and flipped classroom without their knowledge at the beginning of study. Each batch of participants, ranging from year 1 to year 3 will have two groups of study.

Subjects:

Physiotherapy Students. participants from each intake will be randomly allocated into TC(traditional classroom) and FC(flipped classroom).

Inclusion Criteria:

- All physiotherapy participants of University Tunku Abdul Rahman

Exclusion Criteria:

- Participants who are not UTAR physiotherapy participants

Instruments:

Demographic profile of participants Index Of Learning Styles Questionnaire Perception and satisfaction questionnaire Examinations on post teaching session/experiment

Procedures of study:

Study Settings:

Lecture rooms of University Tunku Abdul Rahman Sg. Long Campus.

Sampling Method and Recruitment of Participants:

The number of participants of physiotherapy will first be obtained from the Faculty General Office (FGO) UTAR. Then the participants selected will be grouped into two groups of traditional classroom (TC) and Flipped classroom (FC). Since it is a single blinded study, the participants will not know which group they belong to.

Procedures:

The study will be conducted in two phases:

Phase 1

* Perception and Satisfaction questionnaire will be developed
* A validation test will be conducted on the Perception and Satisfaction questionnaire (face, content and construct) before conducting the study. The validation process will involve the participation of lecturers, professors and students by convenience sampling.

Phase 2

* To prevent bias from the researchers, each participant will be given their code as their identification number. Then the participants will be randomly divided into two groups. They will be briefed on the purpose of study (stating that, the investigators would like to see the efficacy of various teaching methods on students' knowledge gain) and procedure of the study (examinations will be conducted, surveys at the end of each class session and at the end of the study). They are requested to fill up basic demographic data, consent form and ILS questionnaire(measuring the learning style of student) before beginning the study.
* In this study, the lecture will be given by the 'Researcher 1' to standardize the input to the participants of the two groups. This will produce a standardized input to the students of the two groups of teaching method.
* For the FC (flipped classroom) group, the length of the pre-recorded lecture videos will be the same which the participants can view it unlimitedly. An assignment will be given for FC group that will be attempted during the discussion class(2 hours) a week after with the lecturer. No grades will be given for the assignment.
* Meanwhile for the TC(traditional classroom) group, a standard lecture class of 1 hour and 1 hour of tutorial class will be conducted on the same topic. The same ungraded assignment will also be given to this group a week after the lecture class to be attempted in the tutorial class
* For the assignment given, a case study on the topic taught will be designed.
* One day gap will be given following the discussion and tutorial class for FC and TC groups respectively following which an examination of 1 hour duration will be conducted to test on their level of knowledge (assessed by exam score) on the topic being taught for both the groups using the same set of questions. The examination papers will be coded and will be marked by the content expert.
* At the end of the study, each participant will be given a feedback questionnaire to evaluate their perception and satisfaction on the teaching method applied on them using the 'Perception and Satisfaction Questionnaire'.

ELIGIBILITY:
Inclusion Criteria:

* All physiotherapy participants of University Tunku Abdul Rahman

Exclusion Criteria:

* Participants who are not UTAR physiotherapy participants

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Exam result | one week
  A paper based exam will be conducted with objective and subjective questions. It will be a 30 mark paper, 15 mark allotted for lower order thinking (knowledge and comprehension) and 15 marks allotted for higher order thinking of application and analysis. This exam will be able to detect one of the component of knowledge gain of student. Therefore Students' level of knowledge will be assessed by exam score.
Perception and satisfaction questionnaire | one week
  This questionnaire comprise of 24 questions, which will measure the perception and satisfaction level of student. Measuring the perception and satisfaction of student, one will be able to measure one of the component of knowledge gain of student. It will comprise of both qualitative and quantitative analysis of the questionnaire. The questionnaire is subdivided into categories (teaching method, time spend in learning, knowledge gain and application, language and communication, satisfaction and motivation) checking all domains of perception and satisfaction. The questionnaire is self developed and is validated before conducting the study.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Parai, MPT, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia